CLINICAL TRIAL: NCT07261891
Title: Ex Vivo Evaluation of JAK-inhibitor and Gene Therapeutical Approach in JAK-STAT Related Disorders (JAKarta Study)
Brief Title: Ex Vivo Evaluation of JAK-inhibitor and Gene Therapeutical Approach in JAK-STAT Related Disorders
Acronym: JAKarta
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: prof. dr. Rik Schrijvers (Other)
Collaborators: Research Foundation - Flanders (Fonds Wetenschappelijk Onderzoek) (Other)
Responsible Party: Sponsor-Investigator, prof. dr. Rik Schrijvers, Prof. dr., Universitaire Ziekenhuizen KU Leuven
Organization: Universitaire Ziekenhuizen KU Leuven (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S69751; G054022N (Other Grant/Funding Number: Fonds Wetenschapelijk Onderzoek Flanders (FWO))
Record Dates: First submitted 2025-06-25; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Primary Immunodeficiency Diseases (PID)
Keywords: JAK inhibitors; STAT1 gain-of-function; gene therapy
MeSH Terms: conditions — Primary Immunodeficiency Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: This is a parallel assignment study with two arms: (1) patients diagnosed with [rare disease] who will receive [describe treatment] and have blood drawn at specific time points, and (2) healthy controls who will undergo matched blood sampling for comparative analysis. Healthy controls will not receive the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients with a monogenic IEI with an hyperactive JAK-STAT pathway (Other): Adult patients presenting with a genetically confirmed or highly suspected disorder leading to an exagerated JAK-STAT pathway.
  Interventions: Diagnostic Test: blood sampling
- Healthy controls (Other): Healthy controls (without immune-mediated disease)
  Interventions: Diagnostic Test: blood sampling

INTERVENTIONS:
Diagnostic Test: blood sampling — Blood/serum samples will be collected during routine clinical visits at the time of planned peripheral venous blood sampling. Samples will be processed and either used immediately (flow cytometry-based cell sorting, gDNA extraction, in vitro functional assays, primary cell culture or single-cell applications) or stored for later analysis.

SUMMARY:
The investigators want to study the JAK-inhibitors and their impact on the immune system and evaluate the potential of a gene-therapeutic strategy

DETAILED DESCRIPTION:
The investigators want to study ex vivo the effect of JAK-inhibitors on the transcriptional profile and immune cell landscape in patients with inborn errors of the JAK-STAT pathway and the ex vivo evaluation of the feasibility of a gene therapeutic approach for STAT1 GOF. Following aspects will be compared:

* To study pSTAT, transcriptional profile and cytokine production on bulk and sorted peripheral blood cell populations following stimulation in the presence or absence of different jakinibs
* To evaluate to what extent jakinibs can normalize the transcriptional in different cell types (or not and identify blind spots of this treatment strategy)
* To evaluate ex vivo the impact of a gene therapeutic approach for STAT1 GOF.

ELIGIBILITY:
Inclusion Criteria:

* Cases (A): adult patients presenting with a genetically confirmed or highly suspected disorder leading to an exagerated JAK-STAT pathway.
* Controls (B): participants eligible for inclusion in this study must fall in one of the following categories:
* Healthy controls (without immune-mediated disease)

Exclusion Criteria:

* Children (< 18 years at time of recruitment)
* Persons unable or unwilling to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in STAT phosphorylation levels in peripheral blood mononuclear cells (PBMCs) after cytokine stimulation with and without JAK inhibitor exposure | From time of inclusion to 24 months
  Quantification via Median fluorescence intensity (MFI) of phosphorylated STAT1, STAT3, and STAT5 using multiparameter flow cytometry in bulk PBMCs and sorted T cells, B cells, NK cells, and monocyte subsets after standardized cytokine stimulation (e.g., IFNα, IFNγ, IL-6, IL-2) with or without JAK inhibitor exposure. Outcomes reported as fold-change relative to baseline.
Change in transcriptional profiles of immune cell subsets during JAK inhibitor treatment | From time of inclusion to 24 months
  Differential gene expression assessed by single-cell RNA sequencing of PBMCs. Outcome is reported as the number of differentially expressed genes (adjusted p<0.05) at different sampling timepoints (n=3)
Impact of ex vivo gene therapeutic correction in STAT1 gain-of-function patient-derived PBMCs | 24 months from inclusion
  On-target editing efficiency measured as percentage of corrected alleles by targeted sequencing.

SECONDARY OUTCOMES:
Mutation-specific differences in response to JAK inhibitor treatment | From time of inclusion to 24 months
  Comparison of cytokine-induced phosphorylation (MFI of pSTAT1, pSTAT3, pSTAT5) and transcriptional responses (differential expression and pathway enrichment) between patients harboring distinct STAT1 gain-of-function variants. Outcomes reported as half-inhibitory concentration IC50 and area under the curve AUC in comparison to baseline
Impact of our gene therapeutic approach on cell viability | From time of inclusion to 24 months
  Cell viability will be measured with MTT-assay
Off target events in our ex vivo gene therapeutic approach | 24 months
  Off-target events detected by GUIDE-seq and confirmed by amplicon sequencing.
Transcriptional correction of our ex vivo gene therapeutic approach | 24 months
  Transcriptional correction measured by single-cell RNA sequencing (fold-change of interferon pathway gene expression).
Functional differentiation capacity of gene therapy-corrected cells | 24 months
  Functional differentiation capacity of corrected cells assessed by flow cytometry (percentages of T, B, NK, and monocyte subsets).

CONTACTS AND LOCATIONS:
Overall Officials: Rik Schrijvers, MD, PhD, Principal Investigator — UZ Leuven
Locations (1):
- University Hospitals Leuven,, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Staels F, Roosens W, Giovannozzi S, Moens L, Bogaert J, Iglesias-Herrero C, Gijsbers R, Bossuyt X, Frans G, Liston A, Humblet-Baron S, Meyts I, Van Aelst L, Schrijvers R. Case report: Myocarditis in congenital STAT1 gain-of function. Front Immunol. 2023 Mar 20;14:1095595. doi: 10.3389/fimmu.2023.1095595. eCollection 2023. PMID 37020552
- [Background] Giovannozzi S, Demeulemeester J, Schrijvers R, Gijsbers R. Transcriptional Profiling of STAT1 Gain-of-Function Reveals Common and Mutation-Specific Fingerprints. Front Immunol. 2021 Feb 17;12:632997. doi: 10.3389/fimmu.2021.632997. eCollection 2021. PMID 33679782
- [Background] Giovannozzi S, Lemmens V, Hendrix J, Gijsbers R, Schrijvers R. Live Cell Imaging Demonstrates Multiple Routes Toward a STAT1 Gain-of-Function Phenotype. Front Immunol. 2020 Jun 9;11:1114. doi: 10.3389/fimmu.2020.01114. eCollection 2020. PMID 32582194